CLINICAL TRIAL: NCT03166956
Title: The Effect of Enteral Glutamine and Vitamin C Supplementation on Interleukin-6 and Clinical Outcomes in Surgical Intensive Care Unit Patients: A Prospective, Double-Blind, Randomized Controlled Trial
Brief Title: Effect of Glutamine and Vitamin C on Interleukin-6 and Clinical Outcomes in Surgical Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Frank Lin, MD, PhD, Department Chairman, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CS#12181
Record Dates: First submitted 2017-05-11; First posted 2017-05-25 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Critical Care
Keywords: Vitamin C; Glutamine; Interleukin-6; Clinical outcomes
MeSH Terms: interventions — Glutamine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a prospective double-blind randomized study for surgical ICU patients whom can sustain enteral feeding. The test group was provided with glutamine and vitamin C (the GA group); the control (C) group was provided with maltodextrin of equivalent calories as that provided in the GA group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA (glutamine and vitamin C) group (Experimental): Interventions of glutamine and vitamin C enteral supplementations were given to surgical intensive care unit (ICU) patients.
  Subjects in the GA group received enteral supplement of 10 g L-glutamine and 90 mg vitamin C per serving provided by Nutritec-Enjoy Nutrition Inc. (Taipei, Taiwan).
  Interventions: Dietary Supplement: Glutamine and vitamin C enteral supplement
- Control (C) group (Placebo Comparator): Placebo:
  Subjects in the C group received isocaloric maltodextrin as placebo.
  Interventions: Dietary Supplement: Glutamine and vitamin C enteral supplement

INTERVENTIONS:
Dietary Supplement: Glutamine and vitamin C enteral supplement — Subjects in the GA group received enteral supplement of 10 g L-glutamine and 90 mg vitamin C per serving provided by Nutritec-Enjoy Nutrition Inc. (Taipei, Taiwan). Subjects in the C group received isocaloric maltodextrin as placebo.

SUMMARY:
Background & Aims. Glutamine is a conditional essential amino acid that was found in reduced plasma amount in Intensive Care Unit (ICU) patients. The supplementations of glutamine and vitamin C potentially have beneficial effects on wound healing and a reduction in infection rate. In this investigation, enteral glutamine and vitamin C were provided for ICU patient, and the associated changes in proinflammatory cytokines and clinical outcomes were investigated.

DETAILED DESCRIPTION:
Background & Aims. Glutamine is a conditional essential amino acid that was found in reduced plasma amount in Intensive Care Unit (ICU) patients. The supplementation of glutamine in ICU patients has been under much debate. Another nutritional supplement, vitamin C, had a beneficial effect on wound healing and a reduction in infection rate. In this investigation, enteral glutamine and vitamin C were provided for ICU patient, and the associated changes in proinflammatory cytokines and clinical outcomes were investigated.

Methods. This is a prospective double-blind randomized study for surgical ICU patients whom can sustain enteral feeding. The test group was provided with glutamine and vitamin C (the GA group); the control (C) group was provided with maltodextrin of equivalent calories as that provided in the GA group. Plasma glutamine, interleukin-6 (IL-6), and clinical data were collected and analyzed with biostatistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 20 and 85 years
* Not enrolled in other clinical trials in the previous 1 month and during the study period
* Surgical ICU patients cared by the 9 participating surgeons

Exclusion Criteria:

* Older than age 85 years
* Pregnant women
* With an abnormal liver function (receiving drugs or clinical therapies)
* Abnormal renal function (under hemodialysis)
* Multiple organ failure (more than 2 organs)
* Expected ICU stay of less than 72 hours

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 | Blood samples were collected for biochemical analyses on the starting day of enteral feeding (day of enrollment), and every 7 days until day of discharge from ICU, or on the day of discharge from ICU, which ever is shorter, assessed up to 14 days.
  Blood samples were collected for biochemical on the starting day of enteral feeding, and every 7 days or on the day of discharge from ICU.
Interleukin-10 | Blood samples were collected for biochemical analyses on the starting day of enteral feeding (day of enrollment), and every 7 days until day of discharge from ICU, or on the day of discharge from ICU, which ever is shorter, assessed up to 14 days.
  Blood samples were collected for biochemical on the starting day of enteral feeding, and every 7 days or on the day of discharge from ICU.
Body mass index (BMI) | At enrollment.
  body height and weight were taken and body mass index (BMI) calculated at baseline.
Acute Physiology and Chronic Health Evaluation II (APACHE II) score | At enrollment.
  APACHE II score was calculated to classify the disease severity.
Plasma glutamine | Blood samples were collected for biochemical analyses on the starting day of enteral feeding, and every 7 days or on the day of discharge from ICU, assessed up to 14 days.
  Blood was collected for analyses of plasma glutamine levels
Red blood cells | On the starting day of enteral feeding (enrollment), and every 7 days or on the day of discharge from ICU, assessed up to 14 days.
  Blood was collected for hematological analyses
Hemoglobin | On the starting day of enteral feeding (enrollment), and every 7 days or on the day of discharge from ICU, assessed up to 14 days.
  Blood was collected for hematological analyses
White blood cells | On the starting day of enteral feeding (enrollment), and every 7 days or on the day of discharge from ICU, assessed up to 14 days.
  Hematological analyses
C reactive protein | On the starting day of enteral feeding (enrollment), and every 7 days or on the day of discharge from ICU, assessed up to 14 days.
  Hematological analyses

SECONDARY OUTCOMES:
Length of hospital stay | Up to one year
  Clinical outcome
Length of ICU stay | Up to one year
  Clinical outcome
Duration of ventilator use | Up to one year
  Clinical outcome
ICU infectious complications | Up to one year
  Clinical outcome
Mortality in ICU stay | Up to one year
  Clinical outcome
Mortality in hospital stay | Up to one year
  Clinical outcome

IPD SHARING:
Plan to Share IPD: No